CLINICAL TRIAL: NCT00644501
Title: Open Label Study to Evaluate Long Term Treatment Effect of DiaPep277® in Patients Who Have Completed Studies 461* (Phase II) or 901** (Pase III)
Brief Title: Long-Term Treatment Effect of DiaPep277 in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Andromeda Biotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 910
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; beta cells; immunomodulation; immunointervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: DiaPep277

INTERVENTIONS:
Drug: DiaPep277 — 1.0mg dose, injected subcutaneously at baseline and every 3 months thereafter (at 0, 3, 6, 9, 12, 15, 18, 21 months)for a total of 8 administrations.

SUMMARY:
The study is an open-label extension study, offering patients who participated and completed previous study 901 to continue treatment with DiaPep277 and clinical follow-up, for 2 additional years. The expectation is first to demonstrate that extended treatment with DiaPep277 is safe and second to evaluate the long-term effectiveness of treatment. Only patients who completed the previous 2-year study and still have beta-cell function above a threshold level will be eligible for this extension study.

ELIGIBILITY:
Inclusion Criteria:

* A patient that participated in previous 461/PO and 901 studies and received all doses of study medication, per protocol.
* Evidence of clinically significant residual beta-cell function demonstrated by MMTT stimulated C-peptide concentrations ≥ 0.20 nmol/L.

Exclusion Criteria:

* The patient is pregnant or intends to become pregnant or is unwilling to use effective contraceptive method throughout the study.
* The subject has clinical evidence of any diabetes-related complication, or severe allergy or immune deficiency.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2008-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Preservation of endogenous insulin secretion/beta-cell function, as measured by mixed-meal tolerance test stimulated C-peptide secretion. | every 6 months up to 24 months from T0

SECONDARY OUTCOMES:
improved metabolic control and the insulin dose required to maintain it. | every 3 months up to 24 months from T0

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Hadassah Medical Organization
Locations (3):
- Israel (3):
  - Wolfson Medical Centre, Holon
  - Diabetic Unit, Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Centre, Petah Tikva